CLINICAL TRIAL: NCT06158854
Title: An Open-Label Phase 1/2 Study Evaluating the Safety and Efficacy of Etentamig (ABBV-383) in AL Amyloidosis
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events (AE)s in Adult Participants With Immunoglobulin Light Chain (AL) Amyloidosis Receiving Etentamig (ABBV-383) as an Intravenous (IV) Infusion
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-209; 2023-503429-20-00 (Other: EU CT)
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Immunoglobulin Light Chain (AL) Amyloidosis
Keywords: Immunoglobulin Light Chain (AL) Amyloidosis; ABBV-383; TNB-383B
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dose Escalation: ABBV-383 (etentamig) Dose A (Experimental): Participants will receive ABBV-383 (etentamig) dose A during the approximately 2 year study duration.
  Interventions: Drug: ABBV-383 (Etentamig)
- Dose Escalation: ABBV-383 (etentamig) Dose B (Experimental): Participants will receive ABBV-383 (etentamig) dose B during the approximately 2 year study duration.
  Interventions: Drug: ABBV-383 (Etentamig)
- Dose Escalation: ABBV-383 (etentamig) Dose C (Experimental): Participants will receive ABBV-383 (etentamig) dose C during the approximately 2 year study duration.
  Interventions: Drug: ABBV-383 (Etentamig)
- Dose Expansion: ABBV-383 (etentamig) (Experimental): Participants will receive ABBV-383 (etentamig) expansion dose B during the approximately 2 year study duration.
  Interventions: Drug: ABBV-383 (Etentamig)

INTERVENTIONS:
Drug: ABBV-383 (Etentamig) — Intravenous Infusion
  Other Names: TNB-383B

SUMMARY:
Immunoglobulin light chain (AL) amyloidosis is the most common form of systemic amyloidosis. AL amyloidosis has many root causes and is characterized by the overproduction of AL that are secreted by clonal bone marrow plasma cells. This is a study to determine adverse events and change in disease activity in adult participants with AL amyloidosis treated with ABBV-383.

Etentamig (ABBV-383) is an investigational drug being developed for the treatment of AL amyloidosis. This study in broken into 2 parts (dose escalation and dose expansion) with 4 arms. During dose escalation (arms 1-3) participants will receive 1 of 3 doses of ABBV-383 to determine the part 2 dose. After completion of the dose escalation portion of the study, the dose expansion (part 2) portion of the study will begin. One arm (arm 4) will begin and participants will receive a dose determined during the dose escalation portion (part 1). Around 76 adult participants with relapsed/refractory AL amyloidosis will be enrolled at approximately 25 sites across the world.

Participants will receive Etentamig (ABBV-383) as an infusion into the vein for up to approximately 2 year study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary systemic immunoglobulin light chain (AL) amyloidosis.
* Eastern Cooperative Oncology Group (ECOG) performance status of <= 2.
* Have at least 1 organ historically impacted by AL amyloidosis.
* Considered AL amyloidosis cardiac risk stage 1, 2, or 3a, or considered risk stage 3b with stable cardiac function and markers for 3 months prior to dosing, and have measurable disease of AL amyloidosis as defined by difference between involved and uninvolved free light chains (dFLC) >= 50 mg/L or meeting high-risk dFLC progression criteria after immediate prior line of therapy.
* Has previously been exposed to a proteasome inhibitor (PI) and an anti-CD38 monoclonal antibody.

Exclusion Criteria:

* Known history of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months.
* Known allergic reaction, significant sensitivity, or intolerance to constituents of the study treatment (and excipients) and/or other products in the same class.
* Participant has the following conditions:

  * Other non-AL amyloid disease;
  * Previous or current diagnosis of symptomatic multiple myeloma (MM), including the presence of lytic bone disease, plasmacytomas, >= 60% plasma cells in the bone marrow, or hypercalcemia (defined as corrected calcium > 11 mg/dL);
  * Active plasma cell leukemia (i.e., either 20% of peripheral white blood cells or > 2.0 × 109/L circulating plasma cells by standard differential);
  * Waldenström's macroglobulinemia;
  * Acute diffuse infiltrative pneumopathy;
  * Major surgery within 28 days prior first dose or planned during study participation;
  * History of organ transplant requiring continued use of immunosuppressants;
  * Acute infections within 14 days prior first dose requiring parenteral therapy (antibiotic, antifungal, or antiviral);
  * Participant has received an autologous stem cell transplant (SCT) within 12 weeks or an allogeneic SCT within 1 year of the first dose of study treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Only: Number of Participants with Dose-Limiting Toxicities (DLT) | Up to 28 Days
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Dose Expansion Only: Percentage of Participants who Achieve Hematologic Complete Response (CR) | Up to 4 years
  Hematologic CR is defined as the percentage of participants who achieve normalization of free light chain levels, negative serum immunofixation, negative urine immunofixation as determined per the modified International Amyloidosis Consensus Criteria (IACC).
Dose Expansion Only: Number of Participants with DLTs | Up to 4 years
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Number of Participants with Adverse Events (AEs) | Up to 4 years
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Hematologic Overall Response Rate (ORR) | Up to 4 Years
  Hematologic ORR is defined as partial response (PR) + very good partial response (VGPR) + complete remission (CR), proportion of participants who achieved a PR or better, per the modified IACC.
Time to Hematologic CR | Up to 4 Years
  Time to hematologic CR is defined as the time from first dose of study drug until CR, per the modified IACC.
Duration of Hematologic CR | Up to 4 Years
  Duration of hematologic CR is defined as the time from CR until disease progression, per the modified IACC.
Organ Response Rate (OrRR) | Up to 4 Years
  Organ response rate is defined as the time from first dose of study drug until to response in the heart kidney and liver, per the IACC.
Time to Organ Response | Up to 4 Years
  Time to organ response is defined as the time from first dose of study drug until organ response, per the IACC.
Dose Escalation Only: Percentage of Participants who Achieve Hematologic CR Rate as Determined | Up to 4 years
  Hematologic CR is defined as the percentage of participants who achieve normalization of free light chain levels, negative serum immunofixation, negative urine immunofixation as determined per the modified International Amyloidosis Consensus Criteria (IACC).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (11):
  - Sylvester Comprehensive Cancer Center - University of Miami /ID# 255856, Miami, Florida
  - Boston Medical Center /ID# 255066, Boston, Massachusetts
  - Mayo Clinic - Rochester /ID# 255258, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai /ID# 255408, New York, New York
  - Columbia University Medical Center /ID# 255068, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 255073, New York, New York
  - Atrium Health Levine Cancer Institute /ID# 255074, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 255851, Winston-Salem, North Carolina
  - Oregon Medical Research Center /ID# 255119, Portland, Oregon
  - University of Washington /ID# 261581, Seattle, Washington
  - Wisconsin Medical Center /ID# 255836, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital /ID# 255200, Westmead, New South Wales
  - Princess Alexandra Hospital /ID# 255202, Woolloongabba, Queensland
  - Box Hill Hospital /ID# 255199, Box Hill, Victoria
- France (2):
  - CHU Limoges - Dupuytren 1 /ID# 255370, Limoges, Franche-Comte
  - CHU Toulouse - Hopital Rangueil /ID# 255377, Toulouse, Haute-Garonne
- Alexandra General Hospital /ID# 255542, Athens, Attica, Greece
- IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 255654, Bologna, Italy
- Japan (3):
  - Nagoya City University Hospital /ID# 256086, Nagoya, Aichi-ken
  - Kumamoto University Hospital /ID# 262579, Kumamoto, Kumamoto
  - Japanese Red Cross Medical Center /ID# 256083, Shibuya-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-209